CLINICAL TRIAL: NCT00889876
Title: Effect of Exercise or Metformin on Nocturnal Blood Pressure and Other Risk Factors for Cardiovascular Disease (CVD) Among Obese Adolescents
Brief Title: Effect of Exercise or Metformin on Nocturnal Blood Pressure and Other Risk Factors for CVD Among Obese Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: hard to recruite, no funding
Sponsor: Maria Sandberg Westerstahl (Other)
Responsible Party: Sponsor-Investigator, Maria Sandberg Westerstahl, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2008-000461-28
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2011-02

CONDITIONS: Cardiovascular Diseases
Keywords: Obesity; Adolescents; Nocturnal blood pressure reduction; Insulin metabolism; Cardiovascular structure and function; Treatment; Exercise; Metformin; Insulin; Blood glucose; Impaired nocturnal blood pressure reduction
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Motor Activity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental)
  Interventions: Drug: Metformin group
- Exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Drug: Metformin group — 2000 mg/day for one year
  Arms: Metformin
Behavioral: Exercise — 3 times/week with a personal coach for one year. Endurance training.
  Arms: Exercise

SUMMARY:
The objective is to, among obese adolescents, study impact of regular physical activity or metformin therapy on nocturnal blood pressure and related cardiovascular disease risk factors.

DETAILED DESCRIPTION:
Forty subjects will be assigned to the exercise intervention group, thirty to the metformin therapy group and thirty to the control group. Group I will be treated daily with metformin. Group II will perform exercise (endurance) three times/week with a personal coach and group III will serve as control. All participants will be examined at baseline, after 3 months of intervention, after 6 months of intervention and after one year of intervention. Examination includes anthropometric measures, measures of ambulatory 24-h blood pressure and insulin sensitivity, measures for function and structure of the heart and vessels, analysis of atherogenic factors in the blood, aerobic fitness testing and measurement of daily physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-19 years old at inclusion date
* Obesity according to gender and age specific BMI (Cole 2000)
* Reduced nocturnal systolic blood pressure fall (< 10%)
* Signed informed consent by patient and parents

Exclusion Criteria:

* Cardiovascular disease
* Insulin dependent diabetes mellitus
* Patient on medications that are contraindicated during Metformin treatment
* Pregnancy
* Mental or physical conditions limiting the ability to participate

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2009-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Normalization of nocturnal blood pressure dipping | Before and 3, 6 and 12 months of intervention

SECONDARY OUTCOMES:
Normalization of insulin metabolism and cardiovascular structure and function | Before and 3, 6 and 12 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Claude Marcus, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Karolinska University Hospital Huddinge, Stockholm, Sweden